CLINICAL TRIAL: NCT07082426
Title: EASE Study: Early System Experience With the Abbott Balloon-expandable TAVI System: First-In-Human Study
Brief Title: Early System Experience With the Abbott Balloon-expandable TAVI System: First-In-Human Study
Acronym: EASE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABT-CIP-10542
Record Dates: First submitted 2025-07-14; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: Balloon Expandable TAVI; Transcatheter aortic valve implantation (TAVI); Treatment of patients with symptomatic severe aortic valve stenosis; Aortic stenosis; Cardiovascular disease
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Balloon expandable TAVI (Experimental)
  Interventions: Device: Balloon expandable TAVI

INTERVENTIONS:
Device: Balloon expandable TAVI — Prospective, single-arm, multi-center early experience study.

SUMMARY:
Early System Experience with the Abbott Balloon-expandable TAVI System

DETAILED DESCRIPTION:
The Early System Experience with the Abbott's balloon-expandable TAVI System first-in-human study ('EASE study') will evaluate preliminary clinical evidence on the safety and feasibility of the Abbott's balloon-expandable TAVI system for the treatment of patients with symptomatic severe aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Increased surgical risk
* Appropriate anatomy
* At least 18 years of age
* Willing to return for follow-up assessments

Exclusion Criteria:

* Pregnant or nursing subjects
* Anatomic or comorbid conditions
* Evidence of acute myocardial infarction
* Inoperable/ineligible for surgery
* Renal disease requiring chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Post procedure
  Successful access, delivery of the Abbott BE TAVI valve, and retrieval of the delivery system.
Device success | 30 days
  Intended performance of the valve

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart
Locations (3):
- Georgia (2):
  - Israeli - Georgian Medical Research Clinic Healthycore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
- Republican Centre of Emergency Medicine, Tashkent, Toshknt, Uzbekistan